CLINICAL TRIAL: NCT02636686
Title: An Open-label Extension Study of the Long-term Safety, Tolerability and Efficacy of Drisapersen in Subjects With Duchenne Muscular Dystrophy.
Brief Title: Extension Study of Drisapersen in DMD Subjects
Status: No longer available | Type: Expanded Access
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Other Study IDs: BMN-051-302
Record Dates: First submitted 2015-12-09; First posted 2015-12-22 (Estimated); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: DMD; Duchenne Muscular Dystrophy; Drisapersen; Kyndrisa; exon-skipping; exon-51; BMN-051-302; 051-302
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — PRO051

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: Drisapersen — Subjects will receive 6 mg/kg of drisapersen by subcutaneous injection once weekly. If subjects have experienced an intolerable injection site reaction(s), in consultation with the investigator, the subject may be allowed intermittent injections (8 weeks on/4 weeks off) or weekly intravenous infusions of 3 or 6 mg/kg
  Other Names: PRO051

SUMMARY:
This is a phase IIIb, multi-centre, open-label extension study in male subjects with DMD who previously have been treated with drisapersen, aiming at assessing the safety and efficacy of drisapersen.

DETAILED DESCRIPTION:
This is a phase IIIb, multi-centre, open-label extension study in male subjects with DMD who have previously been treated with drisapersen.

This study aims to enroll up to approximately 220 subjects. The primary dosing arm is drisapersen 6 mg/kg as subcutaneous (SC) injection(s) once a week. All subjects starting with subcutaneous injections will receive a loading dose of twice weekly 6mg/kg drisapersen for the first three weeks of treatment. This study does not have a minimum duration of participation. Subjects will have varying times of study participation depending on when they enter from one of the eligible studies and will be permitted to continue the study until such a time that they withdraw based on protocol-defined criteria, or BioMarin stops the study. Subjects naïve to treatment are not eligible for participation in this study

For subjects who have previously experienced significant safety or tolerability issues in one of the eligible studies, or who experience these during this study, there is the potential of an alternate intermittent dosing arm. This will be agreed in advance with the Medical Monitor.

For subjects who have previously experienced significant injection site reactions in an earlier drisapersen study, or who experience similar reaction(s) during this study, there is the potential to be dosed intravenously.

ELIGIBILITY:
Inclusion Criteria:

1. Any subject who has been previously treated with an exon 51 skipping antisense oligonucleotide (drisapersen or eteplirsen) and is not eligible for another ongoing drisapersen study. Subjects who withdrew from the previous studies due to meeting laboratory safety stopping criteria may be eligible to enroll if:
2. The laboratory parameters that led to stopping have resolved; benefit of further treatment with drisapersen outweighs the risk to the individual subject; and following consultation with the Medical Monitor.
3. Subjects with DMD mutation/deletion within the dystrophin gene and correctable by drisapersen-induced DMD exon 51 skipping.
4. Male subjects age >5 at screening in whom the investigator considers treatment with drisapersen is likely to lead to improvement or prevent worsening of the condition.
5. Continued use of glucocorticoids for a minimum of 60 days prior to study entry with a reasonable expectation that the subject will remain on glucocorticoids for the duration of this study. Changes to or cessation of glucocorticoids will be at the discretion of the investigator conducting this study in consultation with the subject/parent and Medical Monitor.
6. Willing and able to comply with all study requirements and procedures (with the exception of those assessments requiring a subject to be ambulant, for those subjects who have lost ambulation).
7. Able to give informed assent and/or consent in writing by the subject and/or parent(s)/legal guardian (according to local regulations)

Exclusion Criteria:

1. Subjects who have previously been treated with drisapersen and who had a serious adverse experience or who met safety stopping criteria that remains unresolved, which in the opinion of the investigator could have been attributable to drisapersen. Once resolved, subject may be eligible to enter the study following investigator consultation with the Medical Monitor.
2. Use of anticoagulants, anti-thrombotics or antiplatelet agents within 28 days of the first re-dosing of drisapersen. Chronic use of anticoagulants, anti-thrombotics or antiplatelet agents is prohibited during the study. As needed dosing (pro re nata - PRN) may be acceptable (except for aspirin) following discussion with the Medical Monitor.
3. Participation in any investigational clinical trial within 3 months prior to start or during this study (except for other drisapersen studies). If subjects have participated in any other study within the last 6 months this should be discussed with the Medical Monitor prior to start of this study.
4. History of significant medical disorder which may confound the interpretation of safety data (e.g. current or history of renal or liver disease/impairment, history of inflammatory illness)
5. Symptomatic cardiomyopathy. If subject has a left ventricular ejection fraction <45% at start of this study, the investigator should discuss inclusion of subject in this study with the Medical Monitor.
6. A platelet count under the lower limit of normal (LLN) at start of this study. A re-test is possible at a later stage, and if within normal range, the subject may enter the study.

Ages: 5 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Derry Ridgway, MD, Study Director — BioMarin Pharmaceutical
Locations (39):
- Kennedy Krieger Institute, Baltimore, Maryland, United States
- IMAI Research, Buenos Aires, Argentina
- Australia (2):
  - Royal Children's Hosital, Children's Neuroscience Centre, Parkville, Victoria
  - Institute for Neuromuscular Research, Westmead
- Belgium (4):
  - Queen Fabiola Children's University Hospital, Brussels
  - Universitair Ziekenhuis Gent, Afdeling Neurologie, Ghent
  - Universitair Ziekenhuis Gasthuisberg, Leuven
  - Hôpital de La Citadelle, Centre de référence des Maladies, Liège
- MHAT "Alexandrovska, Sofia, Bulgaria
- Czechia (2):
  - Detska Nemocnice, Brno
  - FN Motol, Prague
- France (4):
  - CHU de Nantes - Hôtel Dieu, Nantes
  - Hopital Armand Trousseau, Paris
  - Centre hospitalier de Pau, Pau
  - CHU de Toulouse - Hôpital des Enfants, Toulouse
- Germany (3):
  - Dr. von Haunersches Kinderspital, Bayern, Muenchen
  - Universitaetsklinikum Essen, Essen
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau
- Hadassah, Hebrew University Medical Center, Jerusalem, Israel
- Italy (4):
  - Azienda Universitaria Ospedaliera, Messina
  - IRCCS Ospedale Maggiore Policlinico, Mangiagalli e Regina Elena, Milan
  - IRCCS Ospedale Pediatrico Bambino Gesù, Roma
  - Fondazione IRCCS Policlinico Gemelli, Roma
- Japan (4):
  - Kobe University Hospital, Hyōgo
  - Kumamoto University Hospital, Kumamoto
  - National Hospital Organization, Saitama
  - National Center Hospital of Neurology and Psychiatry, Tokyo
- Netherlands (2):
  - Leiden University Medical Center, Leiden
  - UMCN St. Radboud, Nijmegen
- Oslo Universitetssykehus, Oslo, Norway
- SPCSK Uniwersytet Medyczny w, Warsaw, Poland
- Moscow Pediatrics and Children, Moscow, Russia
- Seoul National University Children's Hospital, Seoul, South Korea
- Spain (3):
  - Hospital Sant Joan de Deu, Barcelona
  - Hospital Infantil La Paz, Madrid
  - Hospital Universitari la Fe, Valencia
- Kaohsiung Medical University Hospital, Kaohsiung City, Taiwan
- Hacettepe Children's Hospsital, Ankara, Turkey (Türkiye)
- UCL Institute of Child Health, London, United Kingdom